CLINICAL TRIAL: NCT04339036
Title: UPCC 04219 Phase 2 Study of Capecitabine-Temozolomide(CapTem) With Yttrium-90 Radioembolization in the Treatment of Patients With Unresectable Metastatic Grade 2/3 Neuroendocrine Tumors
Brief Title: CapTemY90 for Grade 2/3 NET Liver Metastases
Acronym: CapTemY90
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 04219; 04219 (Other: Abramson Cancer Center DOCM); NCT04789109 (obsolete NCT alias)
Record Dates: First submitted 2020-03-30; First posted 2020-04-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Neuroendocrine Tumor Grade 2; Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Capecitabine; Temozolomide; Yttrium-90

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral CapTem + Y90 Radioembolization (Experimental): Capecitabine 750 mg/m2 twice daily orally for 14 days and temozolomide 200 mg/m2 orally on Days 10-14, with 14 days between cycles, to be continued until 1) disease progression or 2) intolerable toxicities.
  Trans-arterial radioembolization (TARE) on Day 7 of cycle 2 and, if needed for the other lobe, Day 7 of either cycle 3 or 4.
  Interventions: Drug: Capecitabine Oral Product; Drug: Temozolomide Oral Product; Combination Product: transarterial radioembolization

INTERVENTIONS:
Drug: Capecitabine Oral Product — Capecitabine 750 mg/m2 twice daily orally for 14 days
  Other Names: Xeloda
Drug: Temozolomide Oral Product — temozolomide 200 mg/m2 orally on Days 10-14, with 14 days between cycles
  Other Names: Temodar
Combination Product: transarterial radioembolization — Trans-arterial radioembolization (TARE) on Day 7 of cycle 2 and, if needed for the other lobe, Day 7 of either cycle 3 or 4.
  Other Names: TARE, y90

SUMMARY:
This is a Phase 2 evaluation of hepatic-progression free survival among patients with Grade 2 liver-dominant NET metastases undergoing combination therapy with CapTem and Y90 radioembolization.The hypothesis is to confirm safety and to assess if disease control is improved relative to expectation from either therapy alone.

A Grade 3 arm was added in 2025.

DETAILED DESCRIPTION:
Patients with liver-dominant Grade 2/3 NET metastases from any primary will start CapTem and undergo simulation angiography for radioembolization planning during the first cycle. If they tolerate CapTem and are not excluded from radioembolization, then TARE will be performed on Day 7 of Cycle 2, with additional TARE of Day 7 of cycle 3 or 4 as needed to treat the entire tumor burden. Patients will remain on CapTem until progression or intolerance.

Primary outcome measure is hepatic progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of histologic grade 2 or 3 well differentiated neuroendocrine tumor with unresectable liver metastases (primary tumor or other extrahepatic disease may be present)
* Patients with at least one measurable liver metastases, with size > 1cm (RECIST criteria)
* Patients with liver dominant disease defined as ≥50% tumor body burden confined to the liver
* Liver tumor burden does not exceed 50% of the liver volume
* Patent main portal vein
* At least 4 weeks since last administration of last chemotherapy and /or radiotherapy
* Age >18 years.
* Life expectancy of greater than 6 months.
* ECOG performance status 0-2.
* Adequate liver function as measured by: Total bilirubin ≤ 2.0mg/dl, ALT, AST ≤5 times ULN, albumin ≥2.5g/dl.
* Patients must have adequate organ and marrow function as defined below:
* platelets >100,000/mcL (may be corrected by transfusion)
* serum creatinine < 2.0 mg/dl
* INR <1.6, (may be corrected by transfusion)
* Ability to understand and the willingness to sign a written informed consent document.
* Women of child bearing potential and fertile men are required to use effective contraception (negative urine or serum βHCG for women of child-bearing age)

Exclusion Criteria:

* Contraindications to capecitibine or temozolomide
* Contraindicated for both contrast-enhanced MRI and CT
* Patients previously treated with transarterial embolization (with or without chemotherapy) or with radioembolization (Y-90 microspheres)
* Contraindication for radioembolization procedures:
* excessive hepatopulmonary shunt as determined by the investigator
* inability to deliver Y90 microspheres without risk of non-target embolization of extra-hepatic structures
* Subjects consenting to the trial who fail their simulation angiography will be removed from the study and replaced.
* Patients may not be receiving any other investigational agents.
* Absolute contraindication to intravenous iodinated contrast (Hx of significant previous contrast reaction, not mitigated by appropriate pre-medication).
* Choledochoenteric anastomosis, transpapillary stent or sphincterotomy of duodenal papilla;
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and lactating women are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Intra-hepatic progression-free survival | 2 years. Time from initiation of study therapy until first documented intra-hepatic disease progression, death due to any cause or last scan date that documented intra-hepatic progression-free status.
  Intra-hepatic progression-free survival by RECIST 1.0 is defined as the time from initiation of study therapy until first documented intra-hepatic disease progression, death due to any cause or last scan date that documented intra-hepatic progression-free status.

SECONDARY OUTCOMES:
Overall Progression free survival | 2 years. time from initiation of study therapy until first documented intra- or extra-hepatic disease progression, death due to any cause or last scan date that documented progression-free status
  Overall progression-free survival is defined as the time from initiation of study therapy until first documented intra- or extra-hepatic disease progression, death due to any cause or last scan date that documented progression-free status
Intra-hepatic tumor responses by RECIST | 2 years. from time of initiation of study therapy until subject comes off of study, or study closes
  Intra-hepatic tumor responses will be evaluated by RECIST.
Intra-hepatic tumor responses by EASL | 2 years. from time of initiation of study therapy until subject comes off of study, or study closes
  Intra-hepatic tumor responses will be evaluated by EASL criteria.
extra-hepatic tumor responses | 2 years. from time of initiation of study therapy until subject comes off of study, or study closes
  extra-hepatic tumor responses will be evaluated by RECIST.
Number of participants with systemic toxicities | From period of enrollment to 24 months after last treatment
  Systemic toxicities will be individually assessed by NCI CTCAE Version 4.
Number of participants with hepatic toxicities | From period of enrollment to 24 months after last treatment
  Hepatic toxicities will be individually assessed by NCI CTCAE Version 4.
Change in CgA over time | Tumor markers will be assessed at baseline and then every 3 months for 24 months.
  The primary marker is CgA. Additional cancer site-specific (i.e., gastrinoma) markers may also be assayed.
Quality of Life by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Neuroendocrine tumor | Quality of life will be measured at baseline and then every 3 months for 24 months .
  Quality of Life will be measure by a validated NET-specific instrument, EORTC. Scale is 0-100, higher scores indicate worse symptoms/functioning

CONTACTS AND LOCATIONS:
Overall Officials: Michael Soulen, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - UC San Diego, La Jolla, California
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Modlin IM, Moss SF, Chung DC, Jensen RT, Snyderwine E. Priorities for improving the management of gastroenteropancreatic neuroendocrine tumors. J Natl Cancer Inst. 2008 Sep 17;100(18):1282-9. doi: 10.1093/jnci/djn275. Epub 2008 Sep 9. PMID 18780869
- [Background] Norheim I, Oberg K, Theodorsson-Norheim E, Lindgren PG, Lundqvist G, Magnusson A, Wide L, Wilander E. Malignant carcinoid tumors. An analysis of 103 patients with regard to tumor localization, hormone production, and survival. Ann Surg. 1987 Aug;206(2):115-25. doi: 10.1097/00000658-198708000-00001. PMID 2440390
- [Background] Talamonti MS, Stuart K, Yao JC. Neuroendocrine tumors of the gastrointestinal tract: how aggressive should we be? In: Perry M, ed. American Society of Clinical Oncology 2004 Education Book. Alexandria: American Society of Clinical Oncology, 2004;206-215.
- [Background] Arnold R, Trautmann ME, Creutzfeldt W, Benning R, Benning M, Neuhaus C, Jurgensen R, Stein K, Schafer H, Bruns C, Dennler HJ. Somatostatin analogue octreotide and inhibition of tumour growth in metastatic endocrine gastroenteropancreatic tumours. Gut. 1996 Mar;38(3):430-8. doi: 10.1136/gut.38.3.430. PMID 8675099
- [Background] Saltz L, Trochanowski B, Buckley M, Heffernan B, Niedzwiecki D, Tao Y, Kelsen D. Octreotide as an antineoplastic agent in the treatment of functional and nonfunctional neuroendocrine tumors. Cancer. 1993 Jul 1;72(1):244-8. doi: 10.1002/1097-0142(19930701)72:13.0.co;2-q. PMID 8389666
- [Background] Rinke A, Muller HH, Schade-Brittinger C, Klose KJ, Barth P, Wied M, Mayer C, Aminossadati B, Pape UF, Blaker M, Harder J, Arnold C, Gress T, Arnold R; PROMID Study Group. Placebo-controlled, double-blind, prospective, randomized study on the effect of octreotide LAR in the control of tumor growth in patients with metastatic neuroendocrine midgut tumors: a report from the PROMID Study Group. J Clin Oncol. 2009 Oct 1;27(28):4656-63. doi: 10.1200/JCO.2009.22.8510. Epub 2009 Aug 24. PMID 19704057
- [Background] Caplin ME, Pavel M, Cwikla JB, Phan AT, Raderer M, Sedlackova E, Cadiot G, Wolin EM, Capdevila J, Wall L, Rindi G, Langley A, Martinez S, Blumberg J, Ruszniewski P; CLARINET Investigators. Lanreotide in metastatic enteropancreatic neuroendocrine tumors. N Engl J Med. 2014 Jul 17;371(3):224-33. doi: 10.1056/NEJMoa1316158. PMID 25014687
- [Background] Yao JC, Shah MH, Ito T, Bohas CL, Wolin EM, Van Cutsem E, Hobday TJ, Okusaka T, Capdevila J, de Vries EG, Tomassetti P, Pavel ME, Hoosen S, Haas T, Lincy J, Lebwohl D, Oberg K; RAD001 in Advanced Neuroendocrine Tumors, Third Trial (RADIANT-3) Study Group. Everolimus for advanced pancreatic neuroendocrine tumors. N Engl J Med. 2011 Feb 10;364(6):514-23. doi: 10.1056/NEJMoa1009290. PMID 21306238
- [Background] Raymond E, Dahan L, Raoul JL, Bang YJ, Borbath I, Lombard-Bohas C, Valle J, Metrakos P, Smith D, Vinik A, Chen JS, Horsch D, Hammel P, Wiedenmann B, Van Cutsem E, Patyna S, Lu DR, Blanckmeister C, Chao R, Ruszniewski P. Sunitinib malate for the treatment of pancreatic neuroendocrine tumors. N Engl J Med. 2011 Feb 10;364(6):501-13. doi: 10.1056/NEJMoa1003825. PMID 21306237
- [Background] Gaba RC. Chemoembolization practice patterns and technical methods among interventional radiologists: results of an online survey. AJR Am J Roentgenol. 2012 Mar;198(3):692-9. doi: 10.2214/AJR.11.7066. PMID 22358011
- [Background] Kennedy AS, Dezarn WA, McNeillie P, Coldwell D, Nutting C, Carter D, Murthy R, Rose S, Warner RR, Liu D, Palmedo H, Overton C, Jones B, Salem R. Radioembolization for unresectable neuroendocrine hepatic metastases using resin 90Y-microspheres: early results in 148 patients. Am J Clin Oncol. 2008 Jun;31(3):271-9. doi: 10.1097/COC.0b013e31815e4557. PMID 18525307
- [Background] Saxena A, Chua TC, Bester L, Kokandi A, Morris DL. Factors predicting response and survival after yttrium-90 radioembolization of unresectable neuroendocrine tumor liver metastases: a critical appraisal of 48 cases. Ann Surg. 2010 May;251(5):910-6. doi: 10.1097/SLA.0b013e3181d3d24a. PMID 20395859
- [Background] Memon K, Lewandowski RJ, Mulcahy MF, Riaz A, Ryu RK, Sato KT, Gupta R, Nikolaidis P, Miller FH, Yaghmai V, Gates VL, Atassi B, Newman S, Omary RA, Benson AB 3rd, Salem R. Radioembolization for neuroendocrine liver metastases: safety, imaging, and long-term outcomes. Int J Radiat Oncol Biol Phys. 2012 Jul 1;83(3):887-94. doi: 10.1016/j.ijrobp.2011.07.041. Epub 2011 Dec 2. PMID 22137020
- [Background] Pavel M, Baudin E, Couvelard A, Krenning E, Oberg K, Steinmuller T, Anlauf M, Wiedenmann B, Salazar R; Barcelona Consensus Conference participants. ENETS Consensus Guidelines for the management of patients with liver and other distant metastases from neuroendocrine neoplasms of foregut, midgut, hindgut, and unknown primary. Neuroendocrinology. 2012;95(2):157-76. doi: 10.1159/000335597. Epub 2012 Feb 15. No abstract available. PMID 22262022
- [Background] Strosberg JR, Fine RL, Choi J, Nasir A, Coppola D, Chen DT, Helm J, Kvols L. First-line chemotherapy with capecitabine and temozolomide in patients with metastatic pancreatic endocrine carcinomas. Cancer. 2011 Jan 15;117(2):268-75. doi: 10.1002/cncr.25425. Epub 2010 Sep 7. PMID 20824724
- [Background] Fine RL, Gulati AP, Krantz BA, Moss RA, Schreibman S, Tsushima DA, Mowatt KB, Dinnen RD, Mao Y, Stevens PD, Schrope B, Allendorf J, Lee JA, Sherman WH, Chabot JA. Capecitabine and temozolomide (CAPTEM) for metastatic, well-differentiated neuroendocrine cancers: The Pancreas Center at Columbia University experience. Cancer Chemother Pharmacol. 2013 Mar;71(3):663-70. doi: 10.1007/s00280-012-2055-z. Epub 2013 Jan 31. PMID 23370660
- [Background] Cives M, Ghayouri M, Morse B, Brelsford M, Black M, Rizzo A, Meeker A, Strosberg J. Analysis of potential response predictors to capecitabine/temozolomide in metastatic pancreatic neuroendocrine tumors. Endocr Relat Cancer. 2016 Sep;23(9):759-67. doi: 10.1530/ERC-16-0147. PMID 27552969
- [Background] Cohen SJ, Konski AA, Putnam S, Ball DS, Meyer JE, Yu JQ, Astsaturov I, Marlow C, Dickens A, Cade DN, Meropol NJ. Phase I study of capecitabine combined with radioembolization using yttrium-90 resin microspheres (SIR-Spheres) in patients with advanced cancer. Br J Cancer. 2014 Jul 15;111(2):265-71. doi: 10.1038/bjc.2014.344. Epub 2014 Jul 1. PMID 24983373
- [Background] Hickey R, Mulcahy MF, Lewandowski RJ, Gates VL, Vouche M, Habib A, Kircher S, Newman S, Nimeiri H, Benson AB, Salem R. Chemoradiation of hepatic malignancies: prospective, phase 1 study of full-dose capecitabine with escalating doses of yttrium-90 radioembolization. Int J Radiat Oncol Biol Phys. 2014 Apr 1;88(5):1025-31. doi: 10.1016/j.ijrobp.2013.12.040. PMID 24661655
- [Background] Vinik E, Carlton CA, Silva MP, Vinik AI. Development of the Norfolk quality of life tool for assessing patients with neuroendocrine tumors. Pancreas. 2009 Apr;38(3):e87-95. doi: 10.1097/MPA.0b013e31819b6441. PMID 19276865
- [Background] Vinik E, Silva MP, Vinik AI. Measuring the relationship of quality of life and health status, including tumor burden, symptoms, and biochemical measures in patients with neuroendocrine tumors. Endocrinol Metab Clin North Am. 2011 Mar;40(1):97-109, viii. doi: 10.1016/j.ecl.2010.12.008. PMID 21349413
- [Background] Yadegarfar G, Friend L, Jones L, Plum LM, Ardill J, Taal B, Larsson G, Jeziorski K, Kwekkeboom D, Ramage JK; EORTC Quality of Life Group. Validation of the EORTC QLQ-GINET21 questionnaire for assessing quality of life of patients with gastrointestinal neuroendocrine tumours. Br J Cancer. 2013 Feb 5;108(2):301-10. doi: 10.1038/bjc.2012.560. Epub 2013 Jan 15. PMID 23322194
- [Background] Soulen MC, van Houten D, Teitelbaum UR, Damjanov N, Cengel KA, Metz DC. Safety and Feasibility of Integrating Yttrium-90 Radioembolization With Capecitabine-Temozolomide for Grade 2 Liver-Dominant Metastatic Neuroendocrine Tumors. Pancreas. 2018 Sep;47(8):980-984. doi: 10.1097/MPA.0000000000001115. PMID 30028446
- [Background] Kunz PL, Graham NT, Catalano PJ, Nimeiri HS, Fisher GA, Longacre TA, Suarez CJ, Martin BA, Yao JC, Kulke MH, Hendifar AE, Shanks JC, Shah MH, Zalupski MM, Schmulbach EL, Reidy-Lagunes DL, Strosberg JR, O'Dwyer PJ, Benson AB 3rd. Randomized Study of Temozolomide or Temozolomide and Capecitabine in Patients With Advanced Pancreatic Neuroendocrine Tumors (ECOG-ACRIN E2211). J Clin Oncol. 2023 Mar 1;41(7):1359-1369. doi: 10.1200/JCO.22.01013. Epub 2022 Oct 19. PMID 36260828